CLINICAL TRIAL: NCT01844609
Title: An English Language Obstetrics and Gynecology Journal Club to Improve Medical English in China: A Randomized Controlled Trial
Brief Title: China Obstetrics and Gynecology Journal Club
Acronym: COG-JOCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: First Affiliated Hospital of Heilongjiang Chinese Medicine University (Other)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 42338
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Language Disorders
Keywords: Comprehension; Verbal Learning; Writing; Testing
MeSH Terms: conditions — Language Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self Study Journal Club (Experimental): 25 Chinese Medical Professionals that will be participating in Self Study Journal Club Meetings three times a week for one hour for 8 weeks with interactive questions and answers and discussion of the journal articles.
  Interventions: Behavioral: Self Study Journal Club
- Intensive Journal Club (Experimental): 25 Chinese Medical Professionals that will be participating Face to Face Journal Club Meetings three times a week for one hour for 8 weeks along with a native English speaking mentor.
  Interventions: Behavioral: Intensive Journal Club

INTERVENTIONS:
Behavioral: Self Study Journal Club — This Self Study Journal Club will read articles and prepare written answers to the study questions on their own time. The participants will read 24 articles; 12 gynecology and 12 obstetrics, based on monthly journal clubs available online at the Obstetrics and Gynecology website. The first and last article will serve as a basis for the oral and written exam in which they will be tested on comprehension, verbal and written Medical English.
  Arms: Self Study Journal Club
Behavioral: Intensive Journal Club — This Intensive Journal Club will read articles and prepare written answers to the study questions along with a fluent English speaker. The participants will read 24 articles; 12 gynecology and 12 obstetrics, based on monthly journal clubs available online at the Obstetrics and Gynecology website. Participants will prepare oral presentations of the studies and answers to the study questions. They will have interactive sessions with this fluent English speaking monitor 3 times a week, one hour sessions for 8 weeks. The first and last article will serve as a basis for the oral and written exam in which they will be tested on comprehension, verbal and written Medical English.
  Arms: Intensive Journal Club

SUMMARY:
The purpose of this study is to determine if an intensive journal club based on articles and materials provided on the journal Obstetrics and Gynecology Website improves written and spoken comprehension of medical English in a population of Chinese medical professionals.

DETAILED DESCRIPTION:
This will be a randomized educational trial of an intensive journal club compared to a self study journal club (1:1 randomization). Randomization will take place after baseline.

The population will consist of 50 medical professionals at Heilongjiang University in Harbin China, who agree to participate in an 8 week educational intervention.

This study will assess the impact of applying English for Specific Purposes(ESP) pedagogy to foreign medical education and specifically evaluate learning in the field of obstetrics and gynecology(Ob-Gyn). ESP is a subdivision of a wider field, Language for Specific Purposes(LSP), defined as the area of inquiry and practice in the development of language programs for people who need a language to meet a predictable range of communicative needs. ESP emphasizes teaching language in context and designs a curriculum around the results of a needs assessment, to more accurately determine which language skills are of priority: listening, reading, speaking, and writing. Part of the theory behind ESP suggests that being able to use the vocabulary and structures that students learn in a meaningful context reinforces what is taught and increases motivation. Further, findings from a study by Okamura (2006) that examined how learners succeed in mastering scientific discourse in English showed that they focused on reading academic texts in their field to learn typical writing patterns. This is as opposed to junior learners who focused on mastering the English language by reading English texts written by authors from a breadth of fields. This application of ESP thus reflects how content-specific source articles could serve as rhetorical models and suggests that source articles are able to mediate scholarly writing and learning within the zone of proximal developmental; that is, learners are simultaneously gaining new content knowledge while increasing their skill base.

The proposed intervention is to design an ESP curriculum for medical professionals, specifically Ob-Gyn physicians and researchers at a Chinese Medical University, based on the journal club format and source articles. The study will quantitatively assess the impact of this model on student's ESP language comprehension as well as determine the necessity of the traditional "facilitator" role for a journal club whose purpose is to foster language literacy in non-English speaking universities.

ELIGIBILITY:
Inclusion Criteria:

* Chinese medical professional

Exclusion Criteria:

* English speaking fluency
* Non-Chinese speaking medical professional

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in score from baseline on a 30 question multiple choice exam (questions and answers will be read to the participants) based on APGO-CREOGH shelf exams. | Baseline to 8 weeks

SECONDARY OUTCOMES:
Change in score from baseline on a written (short answer) exam and on an oral exam. | Baseline to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Legro, M.D., Principal Investigator — Milton S. Hershey Medical Center
Locations (2):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States
- First Affiliated Hospital Heilongjiang University of Chinese Medicine, Harbin, China

REFERENCES:
- [Derived] Tsui IK, Dodson WC, Kunselman AR, Kuang H, Han FJ, Legro RS, Wu XK. Chinese Obstetrics & Gynecology journal club: a randomised controlled trial. BMJ Open. 2016 Jan 28;6(1):e010178. doi: 10.1136/bmjopen-2015-010178. PMID 26823180